CLINICAL TRIAL: NCT06570733
Title: Acceptability Research on Integrated Point of Care Sexually Transmitted Infection (STI) Testing and Expedited Partner Therapy (EPT)
Acronym: ARISE
Status: Active, not recruiting | Type: Observational
Sponsor: Wits RHI Research Centre Clinical Research Site (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Thesla Palanee-Phillips, Director of Clinical Trials, Wits RHI Research Centre Clinical Research Site
Other Study IDs: ARISE
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Neisseria Gonorrhea; Trichomoniasis Vaginalis; Chlamydia Trachomatis Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological specimens such as blood samples and vaginal fluid for use in future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol builds on nearly a decade of collaborative HIV/STI prevention research to conduct a prospective cohort study of Adolescent Girls and Young Women (AGYW) eligible for PrEP in South Africa in which we will assess the acceptability of point-of-care STI testing plus Expedited Partner Therapy (EPT) and its impact on the incidence of common curable STIs over 12 months of follow-up. The social-behavioral scientist will undertake qualitative interviews with participants and their male partners to identify facilitators and barriers to EPT uptake and conduct a comparative cost analysis to estimate the cost per person tested using point-of-care STI testing with and without EPT incremental to the cost of standard of care. Findings from the proposed research will provide essential knowledge for national policymakers to advance approaches to STI screening and treatment that will lead to improvements in AGYW sexual reproductive health and reductions in STIs. The data generated from this project are essential to inform efforts to reduce the burden of STIs and HIV-1 in women and achieve the 2030 Sustainable Development Goals, which includes substantial reductions in HIIV and STIs in key at-risk populations. This project will support global efforts to substantially reduce STIs in key populations.

DETAILED DESCRIPTION:
The study aims to estimate the incidence of STIs (Chlamydia trachomatis, Neisseria gonorrhea, and Trichomoniasis vaginalis) among Adolescent Girls and Young Women (AGYW) initiating PrEP who received point-of-care STI testing plus Expedited Partner Therapy (EPT) and those who received point-of-care STI testing but declined EPT. To assess the acceptability of point-to-care STI testing plus EPT for AGYW initiating oral PrEP and its impact on exposure to social harms. To assess the male partner's response and acceptability among those who received EPT. Estimate the cost of implementing rapid point-of-care diagnostic STI testing and EPT for AGYW in South Africa using PrEP compared to standard syndromic management. The study design aims to conduct a prospective cohort study among adolescent girls and young women (AGYW) and assess the incidence of select STIs detected by point-of-care testing, including C.trachomatis, N. gonorrhea, or T. vaginalis, over 12 months of follow-up. Moreover, to assess the acceptability of expedited partner treatment offered to AGYW with an STI and their partners who received EPT. To conduct a comparative cost analysis to estimate the cost per person tested using point-of-care STI testing with and without EPT incremental to the standard cost.

ELIGIBILITY:
Inclusion Criteria:

1. Cisgender girls and women (16-25 years of age, inclusive)
2. Vaginal sex with a cisgender male partner in the last three months
3. CT, GC, or TV detected at screening
4. Willing to return for quarterly study visits
5. Not currently pregnant and not planning to become pregnant in the next 12 months
6. Using or willing to initiate a highly effective method of contraception*
7. HIV-uninfected
8. Interested in initiating oral PrEP
9. No known contraindications to FTC or TDF

Exclusion Criteria:

1. At Screening or Enrollment, participant reports known adverse reaction to FTC or TDF.
2. At Screening or Enrollment, has single or dual rapid Antibody positive reactive HIV-1 test.
3. At Screening or Enrollment, is already participating in another research study involving drugs, medical devices, or vaccines for STI prevention or treatment.
4. As determined by the PIs/designee, any current or historical physical health, mental health or social issue or condition that the site investigator or designee determines should exclude participation.
5. Has any other condition that, in the opinion of the PIs/designee, would preclude informed consent, make study participation unsafe, or otherwise interfere with achieving the study objectives.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants should be cisgender female.
Study Population: Approximately 400 non-pregnant, HIV-negative, cis-gender AGYW aged 16-25, who have recently initiated oral PrEP or who are interested in initiating oral PrEP and are diagnosed with an STI at screening (C. trachomatis, N. gonorrhoeae, or T. vaginalis).
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
GeneXpert | 2 years
  A PCR instrument used to diagnose chlamydia trachomatis and gonorrhea.

SECONDARY OUTCOMES:
Osom rapid testing kit | 2 years
  A rapid testing kit to diagnose trichomoniasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Wits RHI Research Centre, Hillbrow, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
Participants' study information will not be released without their written permission, except as necessary for review, monitoring, and/or auditing by the following:
  * Representatives of the US Federal Government, the US Office for Human Research Protections, National Institutes of Health (NIH) and/or contractors of the NIH, and other local, US, and international regulatory entities
  * Study staff
  * IRBs/ECs Overall study results will be disseminated and published by the University of Washington.